CLINICAL TRIAL: NCT00944905
Title: A Phase I, Multicenter, Open-Label, Dose-Escalation, Multidose Study of MDX-1203 in Subjects With Advanced/Recurrent Clear Cell Renal Cell Carcinoma or Relapsed/Refractory B-Cell Non Hodgkin's Lymphoma
Brief Title: Study of MDX-1203 in Subjects With Advanced/Recurrent Clear Cell Renal Cell Carcinoma (ccRCC) or Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma (B-NHL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX1203-01; CA211-001 (Other: BMS)
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Renal Cell Carcinoma; Non-hodgkin's Lymphoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Lymphoma, Non-Hodgkin | interventions — MDX-1203

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDX-1203 (Experimental): Accelerated titration design (ATD)of 6 dose levels. Subjects will be assigned to a dose level in the order they enter the study
  Interventions: Biological: MDX-1203

INTERVENTIONS:
Biological: MDX-1203 — Assigned Interventions: Single dose of MDX-1203 will be administered every 21 days as an intravenous (i.v.) infusion. Subjects will receive one dose of MDX-1203.

SUMMARY:
The purpose of this study is to determine if MDX-1203 is safe for the treatment of renal cell carcinoma or non-hodgkin's lymphoma.

DETAILED DESCRIPTION:
Multicenter, open-label, dose-escalation, multidose study of MDX-1203, a fully human monoclonal antibody drug conjugate targeting the CD70 transmembrane cell-surface protein which is highly expressed in ccRCC and B-NHL. MDX-1203 is composed of a human anti-CD70 monoclonal antibody covalently linked to a prodrug form of a cytotoxic deoxyribonucleic acid (DNA) minor-groove binding agent (MGBA).

The study will consist of 3 periods: Screening (up to 28 days), Treatment (up to 17 cycles or 2 years), and Follow-up (up to 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
* Criteria specific to each tumor type:

  * For Clear cell renal cell carcinoma (ccRCC): advanced or recurrent disease. Must have failed at least 1 prior systemic therapy
  * For B-cell non-Hodgkin's lymphoma (B-NHL): Must have failed at least 1 prior systemic therapy
* Measurable disease criteria by tumor type:

  * For ccRCC: At least 1 unidimensional measurable lesion
  * For B-NHL: At least 1 bidimensionally measurable lesion
* Prior therapies for advanced/recurrent ccRCC or relapsed/refractory B-NHL or have become intolerant to a systemic therapy
* Provide archived or fresh tumor tissue for CD70 status. Subjects must be CD70+
* Provision of fresh tissue (pre-treatment and on-treatment) for exploratory analysis is mandatory for at least 5 and a maximum of 10 B-NHL subjects

Exclusion Criteria:

* Prior therapy with an anti-CD70 antibody
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Active or untreated central nervous system lymphoma
* Active infection (viral, bacterial, or fungal)
* Evidence of bleeding diathesis or coagulopathy
* Active autoimmune disease requiring immunosuppressive therapy
* Known current drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety profile of MDX-1203 and determine the maximum tolerated dose (MTD) | up to 17 cycles

SECONDARY OUTCOMES:
Biomarker: Incidence of CD70+ tumors in target population | Screening

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University Winship Cancer Center, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - The University of Michigan Health System, Ann Arbor, Michigan